CLINICAL TRIAL: NCT05651555
Title: Evaluation of the EHPAD Caregiver/Pact & Pad Psycho-educational Program for Caregivers With an Institutionalized Parent
Acronym: EAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP220084; 2021-A00553-38 (Other: France : ANSM)
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Caregivers
Keywords: Caregiving; Psychosocial intervention; Nursing home placement; Nursing home admission; Informal long-term care
MeSH Terms: interventions — Protein-Arginine Deiminases; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N arm (Experimental)
  Interventions: Behavioral: Psycho-educational program EHPAD caregivers / Pact & Pad for caregivers with a parent in an institution
- Control group (Active Comparator)
  Interventions: Behavioral: Psycho-educational program EHPAD caregivers / Pact & Pad for caregivers with a parent in an institution

INTERVENTIONS:
Behavioral: Psycho-educational program EHPAD caregivers / Pact & Pad for caregivers with a parent in an institution — Psycho-educational program EHPAD caregivers / Pact & Pad for caregivers with a parent in an institution

SUMMARY:
Moving into an institution is a new stage in the life of the patient but also of the caregiver. The caregiver is overwhelmed by various feelings such as loss of control, powerlessness, guilt, sadness, the feeling of loneliness at home but also relief. This experience can be characterized by great anxiety and the feeling of being misunderstood by the family and professional environment.

This emotional state is not without consequences for the caregiver/resident and caregiver/care team relationship.

Several factors have been identified that may be at the origin of these states.

A new training, information and support program has been created to present these different factors to caregivers and to allow them to address them with professionals in a group setting.

DETAILED DESCRIPTION:
In 2015, there were 593,005 places for dependent elderly people in institutions in France. The increase in the life expectancy of the population and the decrease in the number of caregivers predicted by the World Health Organization suggests that institutions will be increasingly solicited. Also, due to the increase in neurodegenerative diseases, family caregivers are being forced to resort to institutionalization. According to the study conducted by the number of family caregivers of sick, elderly, or dependent individuals is estimated to be around 11 million in France. 58% of these caregivers are women. 52% work, 86% help a family member, including 41% one of their parents, 34% help several people, compared to 28% in 2017 (multi-caregivers), 57% help a relative in a situation of dependence due to old age (compared to 48% in 2017). Finally, 82% devote at least 20 hours per week on average to their loved one(s), 37% of the caregivers surveyed admit to receiving no outside help even though they are often elderly themselves.

Moving into an institution is a new stage in the life of the patient but also of the caregiver. The caregiver is overwhelmed by various feelings such as loss of control, powerlessness, guilt, sadness, the feeling of loneliness at home but also relief. This experience can be characterized by great anxiety and the feeling of being misunderstood by the family and professional environment.

This emotional state is not without consequences for the caregiver/resident and caregiver/care team relationship.

Several factors have been identified that may be at the origin of these states.

A new training, information and support program has been created to present these different factors to caregivers and to allow them to address them with professionals in a group setting.

Hypothesis 1: The psycho-educational program "EHPAD aidant" containing various information about the financial and medical-psychological care of a resident in an EHPAD, combined with the intervention of various professionals in this sector and a group therapy, allows for a decrease in anxiety symptoms.

Hypothesis 2: The psycho-educational program "EHPAD caregiver" allows for a decrease in depressive symptoms, an improvement in perceived stress, coping strategies, satisfaction, quality of life, the caregiver/caregiver relationship, as well as a decrease in perceived burden and guilt related to the institutionalization of the parent

Hypothesis 3: There is a link between anxiety symptomatology and intolerance of uncertainty.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers defined according to the European charter for family caregivers COFACE: "the non-professional person who comes to the aid mainly, in part or totally, to a person dependent on his or her entourage, for activities of daily living. This regular help can be provided on a permanent basis or not and can take several forms, in particular: nursing, care, support for education and social life, administrative procedures, coordination, permanent vigilance, psychological support, communication, domestic activities. . Currently, these caregivers have an elderly relative living in an institution or in the process of institutionalization
* Have been a caregiver for at least six months
* Have a parent in an EHPAD for less than 25 weeks
* The loved one is not at the end of life when the caregiver starts the program
* Participate in at least five workshops out of the seven offered as part of the program.
* Be of legal age (at least 18 years old)
* Presence of depression or anxiety according to HAD
* Be motivated to follow the program
* Signature of consent.
* Be affiliated with a social security scheme

Exclusion Criteria:

* Caregiver with a loved one living at home without institutionalization plans
* Professional caregivers, former caregivers
* Absence of depression and/or anxiety
* Deceased relative
* Have untreated diagnosed psychiatric disorders
* To be suffering from proven cognitive disorders
* Already benefit from another caregiver assistance program.
* Patient under AME
* Vulnerable people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
HADS (Hospital Anxiety and Depression scale) | Inclusion
  Reduction in anxiety symptoms of 1 to 3 points according to the HADS Hospital Anxiety and Depression scale) between the start and the end of the program.
  The depression score assessed by the HADS will be measured. The maximum score that can be obtained for this sub-score is 21. is possible to determine the presence or not, as well as the intensity of the depressive disorder: absence of depressive disorder (score ranging from 0 to 7), suspected depressive disorder (score ranging from 8 to 10) and proven depressive disorder (score ranging from 11 to 21). Thus, the higher the score, the more severe the participant's symptomatology.
HADS (Hospital Anxiety and Depression scale) | Week 16 for the group N (T2)
  Reduction in anxiety symptoms of 1 to 3 points according to the HADS Hospital Anxiety and Depression scale) between the start and the end of the program.
  The anxiety score assessed by the HADS will be measured. The maximum score that can be obtained for this sub-score is 21. Within the questionnaire, the order of scoring (from 0 to 3 or from 3 to 0) is alternated, in order to limit the bias linked to their repetition. Depending on the participants' scores on the depression subscale, it is possible to determine the presence or not, as well as the intensity of the depressive disorder: absence of depressive disorder (score ranging from 0 to 7), suspected depressive disorder (score ranging from 8 to 10) and proven depressive disorder (score ranging from 11 to 21). Thus, the higher the score, the more severe the participant's symptomatology. The first French validation of this scale was carried out by Lepine et al., 1985.
HADS (Hospital Anxiety and Depression scale) | Week 24 for the group C (T3)
  Reduction in anxiety symptoms of 1 to 3 points according to the HADS Hospital Anxiety and Depression scale) between the start and the end of the program.
  The depression score assessed by the HADS will be measured. The maximum score that can be obtained for this sub-score is 21. Within the questionnaire, the order of scoring (from 0 to 3 or from 3 to 0) is alternated, in order to limit the bias linked to their repetition. Depending on the participants' scores on the depression subscale, it is possible to determine the presence or not, as well as the intensity of the depressive disorder: absence of depressive disorder (score ranging from 0 to 7), suspected depressive disorder (score ranging from 8 to 10) and proven depressive disorder (score ranging from 11 to 21). Thus, the higher the score, the more severe the participant's symptomatology. The first French validation of this scale was carried out by Lepine et al., 1985.

SECONDARY OUTCOMES:
HADS (Hospital Anxiety and Depression scale) | Week 8 (T1) for both groups
  Reduction in anxiety symptoms of 1 to 3 points according to the HADS Hospital Anxiety and Depression scale) between the start and the end of the program.
  The depression score assessed by the HADS will be measured. The maximum score that can be obtained for this sub-score is 21. Within the questionnaire, the order of scoring (from 0 to 3 or from 3 to 0) is alternated, in order to limit the bias linked to their repetition. Depending on the participants' scores on the depression subscale, it is possible to determine the presence or not, as well as the intensity of the depressive disorder: absence of depressive disorder (score ranging from 0 to 7), suspected depressive disorder (score ranging from 8 to 10) and proven depressive disorder (score ranging from 11 to 21). Thus, the higher the score, the more severe the participant's symptomatology. The first French validation of this scale was carried out by Lepine et al., 1985.
HADS (Hospital Anxiety and Depression scale) | Week 16 for the group C (T2)
  Reduction in anxiety symptoms of 1 to 3 points according to the HADS Hospital Anxiety and Depression scale) between the start and the end of the program.
  The depression score assessed by the HADS will be measured. The maximum score that can be obtained for this sub-score is 21. Within the questionnaire, the order of scoring (from 0 to 3 or from 3 to 0) is alternated, in order to limit the bias linked to their repetition. Depending on the participants' scores on the depression subscale, it is possible to determine the presence or not, as well as the intensity of the depressive disorder: absence of depressive disorder (score ranging from 0 to 7), suspected depressive disorder (score ranging from 8 to 10) and proven depressive disorder (score ranging from 11 to 21). Thus, the higher the score, the more severe the participant's symptomatology. The first French validation of this scale was carried out by Lepine et al., 1985.
Zarit Caregiver Burden Scale | Inclusion
  Between 0 and 20 points, the caregiver's burden is considered to be very low or even zero,
  * Between 21 and 40 points, the burden is light,
  * Between 41 and 60 points, the burden is moderate,
  * Between 60 and 88 points, the burden is severe.
Zarit Caregiver Burden Scale | Week 8
  * Between 0 and 20 points, the caregiver's workload is considered to be very low or even zero,
  * Between 21 and 40 points, the burden is light,
  * Between 41 and 60 points, the burden is reduced,
  * Between 60 and 88 points, the burden is severe.
Zarit Caregiver Burden Scale | Week 16
  * Between 0 and 20 points, the caregiver's workload is considered to be very low or even zero,
  * Between 21 and 40 points, the burden is light,
  * Between 41 and 60 points, the burden is reduced,
  * Between 60 and 88 points, the burden is severe.
Zarit Caregiver Burden Scale | Week 24 for the group C (T3)
  * Between 0 and 20 points, the caregiver's workload is considered to be very low or even zero,
  * Between 21 and 40 points, the burden is light,
  * Between 41 and 60 points, the burden is reduced,
  * Between 60 and 88 points, the burden is severe.
CADI (Carers Assessment of Difficulties Index) | Inclusion
  30 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CADI (Carers Assessment of Difficulties Index) | Week 8
  30 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CADI (Carers Assessment of Difficulties Index) | Week 16
  30 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CADI (Carers Assessment of Difficulties Index) | Week 24 for the group C (T3)
  30 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CAMI (Carers Assessment of Managing Index) | Inclusion
  38 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CAMI (Carers Assessment of Managing Index) | Week 8
  38 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CAMI (Carers Assessment of Managing Index) | Week 16
  38 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CAMI (Carers Assessment of Managing Index) | Week 24 for the group C (T3)
  38 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CASI (Carers Assessment of Satisfaction Index) | Inclusion
  30 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CASI (Carers Assessment of Satisfaction Index) | Week 8
  30 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CASI (Carers Assessment of Satisfaction Index) | Week 16
  30 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
CASI (Carers Assessment of Satisfaction Index) | Week 24 for the group C (T3)
  30 items - Rating is done using a three-point scale, ranging from 0: "the proposal does not apply to my situation", to 3: "it is a very stressful difficulty / a very useful strategy/a very great satisfaction"
Quality of life (QOL AD) | Inclusion
  Scoring instructions for QOL-AD:
  Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.
  The total score is the sum of all 13 items
Quality of life (QOL AD) | Week 8
  Scoring instructions for QOL-AD:
  Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.
  The total score is the sum of all 13 items
Quality of life (QOL AD) | Week 16
  Scoring instructions for QOL-AD:
  Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.
  The total score is the sum of all 13 items
Quality of life (QOL AD) | Week 24 for the group C (T3)
  Scoring instructions for QOL-AD:
  Points are assigned to each item as follows: poor = 1, fair = 2, good = 3, excellent = 4.
  The total score is the sum of all 13 items
Visual scale | Inclusion
  Visual scale for the quality of communication caregiver / carers - From 1 (bad quality) to 10 (very good quality).
Visual scale | Week 8
  Visual scale for the quality of communication caregiver / carers - From 1 (bad quality) to 10 (very good quality).
Visual scale | Week 16
  Visual scale for the quality of communication caregiver / carers - From 1 (bad quality) to 10 (very good quality).
Visual scale | Week 24 for the group C (T3)
  Visual scale for the quality of communication caregiver / carers - From 1 (bad quality) to 10 (very good quality).
Visual scale | Inclusion
  Visual scale for the quality of communication caregiver / helped - From 1 (bad quality) to 10 (very good quality).
Visual scale | Week 8
  Visual scale for the quality of communication caregiver / helped - From 1 (bad quality) to 10 (very good quality).
Visual scale | Week 16
  Visual scale for the quality of communication caregiver / helped - From 1 (bad quality) to 10 (very good quality).
Visual scale | Week 24 for the group C (T3)
  Visual scale for the quality of communication caregiver / helped - From 1 (bad quality) to 10 (very good quality).
Scale of Intolerance to Uncertainty | Inclusion
  27 items. Items are rated on a Likert scale from 1 ("Not at all relevant") to 5 ("Completely relevant"). The total score is obtained by adding the items. it will be between 27 and 135 (27*5=135)
Scale of Intolerance to Uncertainty | Week 8
  27 items. Items are rated on a Likert scale from 1 ("Not at all relevant") to 5 ("Completely relevant"). The total score is obtained by adding the items. it will be between 27 and 135 (27*5=135)
Scale of Intolerance to Uncertainty | Week 16
  27 items. Items are rated on a Likert scale from 1 ("Not at all relevant") to 5 ("Completely relevant"). The total score is obtained by adding the items. it will be between 27 and 135 (27*5=135)
Scale of Intolerance to Uncertainty | Week 24 for the group C (T3)
  27 items. Items are rated on a Likert scale from 1 ("Not at all relevant") to 5 ("Completely relevant"). The total score is obtained by adding the items. it will be between 27 and 135 (27*5=135)
Visual scale | Inclusion
  Measure of guilt - From 1 to 10 It assesses the quality of the relationship with the parent in the eyes of the carer (0 = worse outcome / 10 = better outcome).
Visual scale | Week 8
  Measure of guilt - From 1 to 10 It assesses the quality of the relationship with the parent in the eyes of the carer (0 = worse outcome / 10 = better outcome).
Visual scale | Week 16
  Measure of guilt - From 1 to 10 It assesses the quality of the relationship with the parent in the eyes of the carer (0 = worse outcome / 10 = better outcome).
Visual scale | Week 24 for the group C (T3)
  Measure of guilt - From 1 to 10 It assesses the quality of the relationship with the parent in the eyes of the carer (0 = worse outcome / 10 = better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie RIGAUD, MD, PhD, PU-PH, Principal Investigator — Broca Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP)
Locations (1):
- Assistance Publique - Hôpitaux de Paris (AP-HP) - Broca Hospital - Geriatric unit, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meziane-Damnee S, Bayle C, Pino M, Lenoir H, Cantegreil I, Rigaud AS. [A psycho-educational program for family caregivers of people with Alzheimer's disease entering an institution]. Soins Gerontol. 2023 May-Jun;28(161):20-23. doi: 10.1016/j.sger.2023.04.007. Epub 2023 Jun 1. French. PMID 37328202